CLINICAL TRIAL: NCT06175637
Title: Observational Study of the Effectiveness and Safety of the MEK 1/2 Inhibitor (MEKi) Koselugo (Selumetinib) in Pediatric Patients With Symptomatic, Inoperable, Neurofibromatosis Type 1 (NF1)-Associated Plexiform Neurofibromas (PN)
Brief Title: Observational Study to Evaluate the Effect and Safety of Selumetinib in Pediatric Patients With NF1-PNs
Acronym: PEDIA
Status: Active, not recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1346R00016
Record Dates: First submitted 2023-11-08; First posted 2023-12-19 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Neurofibroma, Plexiform
Keywords: Neurofibroma, Plexiform
MeSH Terms: conditions — Neurofibroma, Plexiform

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — No Biospecimen sample will be collected in this study，all participants will receive clinical examination base on routine clinical diagnosis and treatment procedures.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective, multicenter, observational study of Chinese pediatric NF1-PN patients treated with selumetinib. The study will be conducted at approximately 12 centers in China and will include approximately 80-100 patients. Treatment centers that have PN diagnosis and/or selumetinib treatment experience will be targeted for recruitment. Patients/caregivers who are eligible and willing to participate will be enrolled into the study. Patients will start selumetinib treatment after enrollment. The study will have a 16-month enrollment period. Patients will be followed up until the end of a 24-month observation period after first dose of selumetinib, or patient death, lost to follow-up, withdrawal of consent, whichever occurs first. Patients will be followed within a 24-month period (starting after first dose received) in the study even if selumetinib is discontinued. The aims of this study are to expand understanding of disease characteristics and treatment pattern of NF1-PN in China in a real-world setting and to evaluate real-world effectiveness and safety of selumetinib for Chinese pediatric patients with NF1-PN

DETAILED DESCRIPTION:
Neurofibromatosis type 1 (NF1) is a rare and incurable autosomal dominant genetic disorder that is characterized by manifestations in multiple organ systems including tumors of the nervous system. Although NF1 is inherited via autosomal dominance, 50% of detected mutations are de novo. The population prevalence of NF1 estimates ranging from approximately 1/2000 to 1/4000 , and there are estimated 460,000 patients in China. The condition is usually recognized in early childhood, when pigmentary manifestations emerge. NF1 patients have decreased life expectancy of 15 years compared to the general population. High-grade glioma (HGG) and malignant peripheral nerve sheath tumor (MPNST) were noteworthy causes of death among patients with NF1.

Plexiform neurofibromas (PN) are tumors arise from Schwann cells of peripheral, visceral, or subcutaneous nerves, affecting 30%-50% of patients with NF1. PN can cause substantial complications including pain, functional impairment, disfigurement and have a risk of malignant transformation. The lifetime incidence of MPNST in patients with NF1 is 8%-13% , and the presence of a PN elevates the risk of MPNST formation by 20-fold among NF1 patients. Most PN are diagnosed in early childhood and grow most rapidly during this period. Surgical resection is the mainstay treatment for PN, yet surgical treatment does not have satisfactory effect. Complete surgical resection of these tumors is often infeasible due to the extensive growth of the tumor and invasion of surrounding tissues, and partial removal often comes with a high recurrence rate. Conventional chemotherapy and radiotherapy have shown limited efficacy for NF1-associated PN. As a result, medical therapies targeting PN have been evaluated in clinical trials.

The therapeutic revolution came in 2020 with the approval of selumetinib for pediatric patients with NF1-associated PN. Selumetinib is an oral selective inhibitor of MEK 1 and 2 and has been confirmed effective for NF1-associated PN in SPRINT Phase II Stratum 1. The overall response rate was 68% (34/50), and 82% (28/34) of these patients had a durable response (lasting ≥12 months) (Gross AM et al, 2020). Selumetinib was approved by the United States Food and Drug Administration (US-FDA) on April 10, 2020, becoming the first approved targeted therapy for pediatric patients with NF1-associated PN. On April 28, 2023, the China National Medical Products Administration (NMPA) approved selumetinib for pediatric patients aged 3 years and older diagnosed with NF1 who have symptomatic, inoperable PN.

To date, evidence on real-world data of clinical benefit of selumetinib for NF1-associated PN patients among Chinese population is lacking. Moreover, due to the relatively rare affected population, disease knowledge of NF1 and PN is limited among healthcare professionals (HCPs) and throughout the society. An observational study of pediatric patients with NF1-associated PN treated with selumetinib in China will fulfill the data gap of effectiveness and safety of selumetinib for Chinese NF1-PN patients and will facilitate the understanding of disease characteristics and treatment in this population in a real-world setting.

Observational Study of the Effectiveness and Safety of the MEK 1/2 Inhibitor (MEKi) Koselugo (Selumetinib) in Pediatric Patients with Symptomatic, Inoperable, Neurofibromatosis Type 1 (NF1)-Associated Plexiform Neurofibromas (PN) . The aims of this study are to expand understanding of disease characteristics and treatment pattern of NF1-PN in China in a real-world setting and to evaluate real-world effectiveness and safety of selumetinib for Chinese pediatric patients with NF1-PN. This is a prospective, multicenter, observational study of Chinese pediatric NF1-PN patients treated with selumetinib. The study will be conducted at approximately 12 centers in China and will include approximately 80-100 patients (ie, at least 80 patients will be enrolled into the study, but should not enrol more than 100 patients within 16 months). Treatment centers that have PN diagnosis and/or selumetinib treatment experience will be targeted for recruitment. Patients/caregivers who are eligible and willing to participate will be enrolled into the study. Patients will start selumetinib treatment after enrollment.

The study will have a 16-month enrollment period. Patients will be followed up until the end of a 24-month observation period after first dose of selumetinib, or patient death, lost to follow-up, withdrawal of consent, whichever occurs first. Patients will be followed within a 24-month period (starting after first dose received) in the study even if selumetinib is discontinued. Pediatric patients with neurofibromatosis type 1 (NF1) aged 3-16 years (3 and 16 years are inclusive) who have symptomatic, inoperable plexiform neurofibromas (PN) and intend to use selumetinib after enrollment. Approximately 80-100 eligible patients will be enrolled in the study. Exposure to selumetinib is of interest for this study. Based on prescribing information, the recommended dosage of selumetinib is 25 mg/m2 orally twice daily (approximately every 12 hours) until disease progression, unacceptable toxicity, risk or no longer benefit from selumetinib treatment in the judgement of physicians, or the end of 24-month follow-up period, whichever occurs first. After 24-month follow-up period, whether the patients continue exposure to selumetinib will not be collected. Based on the study purpose, the following outcomes will be collected or measured: Patient demographics and disease characteristics at baseline and during selumetinib treatment

Treatment profile with selumetinib

Effectiveness outcomes of selumetinib

Safety outcomes of selumetinib

Time to tumor regrowth after selumetinib discontinuation

Disease and treatment course after selumetinib discontinuation

Caregiver- or patient-reported selumetinib treatment adherence

Patient-reported pain intensity.

ELIGIBILITY:
Inclusion Criteria:

* (1) 3≤ age ≤16 years old at the time of study enrollment; (2) Diagnosed with NF1 as per the revised 2021 Guidelines; (3) Have symptomatic, inoperable PN: (4) Intend to use selumetinib after enrollment; (5) Able to give written informed consent. Data collection must only be done after obtaining written informed consent. Patient or patient's parent/legal guardian must be willing and able to give written informed consent. Parent or legal guardian consent is required in the assent process with appropriate documentation. Mandatory provision of signed and dated parent/legal guardian consent for the study along with the pediatric assent form, when applicable.

Exclusion Criteria:

* (1) Evidence of MPNST, prior malignancy or other cancer requiring treatment with chemotherapy or radiation therapy; (2) A life-threatening illness, medical condition, or organ system dysfunction; (3) Have had prior treatment with a MEKi, Ras or Raf inhibitor; (4) Patients currently participating in any clinical trials at the time of enrollment or initiation of selumetinib.

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The target population of interest in this study is pediatric patients with neurofibromatosis type 1 (NF1) aged 3-16 years (3 and 16 years are inclusive) who have symptomatic, inoperable plexiform neurofibromas (PN) and intend to use selumetinib after enrollment. Each eligible patient should meet all of the inclusion criteria and none of the exclusion criteria. At least 80 and no more than 100 eligible patients will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 409 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
NF1-PN patient demographics and disease characteristics at baseline and during selumetinib treatment | From baseline to 24 months after first dose of selumetinib
  Race,ethnicity,Gender,Date of birth,Relationship of caregiver to patient
NF1-PN disease characteristics | From baseline to 24 months after first dose of selumetinib
  Date of diagnosis or age at diagnosis of NF1, Date of diagnosis or age at diagnosis of PN, NF1 clinical diagnosis criteria and related manifestations, NF1 and PN diagnostic tests and results, Morbidities related to PN
Selumetinib treatment profile | From baseline to 24 months after first dose of selumetinib
  Dose and dose modification, start and stop dates, dose interruption and discontinuation, reasons for interruption, discontinuation and dose modification.
Physician's qualitative assessment of disease status for clinically significant PN and overall disease status | From baseline to 24 months after first dose of selumetinib
  Improving with treatment, progression, stable
NF1 disease status | From baseline to 24 months after first dose of selumetinib
  Presence, number, size (Diameter - centimeters or cubic centimeters of volume) and location (neck/trunk, trunk and limbs, limbs only, head only, head and neck, trunk only) of PN/ optic pathway gliomas/ café-au-lait macules/ cutaneous neurofibroma.

SECONDARY OUTCOMES:
To assess tumor activity of NF1-PN upon discontinuation of selumetinib | From baseline to 24 months after first dose of selumetinib
  Time to tumor regrowth after treatment discontinuation.
To describe the course of patients' disease and treatment following discontinuation of selumetinib | From baseline to 24 months after first dose of selumetinib
  The course of patients' disease and treatment following discontinuation of selumetinib will be analyzed descriptively.
To describe caregiver- or patient-reported treatment adherence | From baseline to 24 months after first dose of selumetinib
  The adherence to treatment will be derived from data collected in the medication diary. Persistence of treatment will be assessed by the time from first dose to discontinuation date and will be analyzed by survival analysis methods.
To determine whether patients treated with selumetinib have a clinically meaningful decrease in pain intensity associated with pain scale | From baseline to 24 months after first dose of selumetinib
  The evolution of pain measured with NRS-11 compared with baseline. Time to pain onset after discontinuation. PROs scales.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Ni, PhD, Principal Investigator — Beijing Children hospital
Locations (25):
- China (25):
  - Research Site, Beijing, Beijing Municipality
  - Research Site, Chongqing, Chongqing Municipality
  - Research Site, Lanzhou, Gansu
  - Research Site, Guangzhou, Guangdong
  - Research Site, Shenzhen, Guangdong
  - Research Site, Nanning, Guangxi
  - Research Site, Guiyang, Guizhou
  - Research Site, Shijiazhuang, Hebei
  - Research Site, Zhengzhou, Henan
  - Research Site, Wuhan, Hubei
  - Research Site, Changsha, Hunan
  - Research Site, Nanjing, Jiangsu
  - Research Site, Suzhou, Jiangsu
  - Research Site, Nanchang, Jiangxi
  - Research Site, Shenyang, Liaoning
  - Research Site, Jinan, Shandong
  - Research Site, Shanghai, Shanghai Municipality
  - Research Site, Taiyuan, Shanxi
  - Research Site, Xi’an, Shanxi
  - Research Site, Chengdu, Sichuan
  - Research Site, Tianjin, Tianjin Municipality
  - Research Site, Kunming, Yunnan
  - Research Site, Hangzhou, Zhejiang
  - Research Site, Wenzhou, Zhejiang
  - Research Site, Nanjing

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal
  Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/